CLINICAL TRIAL: NCT01147757
Title: Effect of Intraoperative Remifentanil Infusion Rate on Postoperative Tolerance and Analgesic Consumption in Pediatric Laparoscopic Ureteroneocystostomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Principal Investigator, Jeong-Yeon Hong, associate professor, Yonsei University
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 4-2010-0129
Record Dates: First submitted 2010-06-17; First posted 2010-06-22 (Estimated); Last update posted 2011-12-06 (Estimated); Status verified 2011-12

CONDITIONS: Pediatrics
Keywords: pediatric patients (ASA physical status I or II) aged between
MeSH Terms: interventions — Remifentanil

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (4):
- saline (Placebo Comparator): Group S (n = 15): saline
  Interventions: Drug: remifentanil
- remifentanil 0.3 mcg/kg/min (Experimental): Group 0.3 (n = 15): remifentanil 0.3 mcg/kg/min
  Interventions: Drug: remifentanil
- remifentanil 0.6 mcg/kg/min (Experimental): Group 0.6 (n = 15): remifentanil 0.6 mcg/kg/min
  Interventions: Drug: remifentanil
- remifentanil 0.9 mcg/kg/min (Experimental): Group 0.9 (n = 15): remifentanil 0.9 mcg/kg/min
  Interventions: Drug: remifentanil

INTERVENTIONS:
Drug: remifentanil — During surgery, 3 different dose of remifentanil or placebo was infused.

SUMMARY:
Effect of intraoperative remifentanil infusion rate on postoperative tolerance and analgesic consumption in pediatric laparoscopic ureteroneocystostomy.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients (ASA physical status I and II) aged between 1-5 yrs and scheduled elective laparoscopic ureteroneocystostomy

Exclusion Criteria:

* cardiovascular, renal, liver disease or growth retardation

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2010-06; Primary Completion 2012-06 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
fentanyl consumption for IV-PCA | 24 h and 48 h after surgery
Postoperative pain score | during 48 h after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Jeong-Yeon Hong, Principal Investigator — Department of Anesthesiology and Pain Medicine, Yonsei University College of Medicine, Seoul, Korea
Locations (1):
- Severance Hospital, Seoul, South Korea